CLINICAL TRIAL: NCT01218308
Title: Efficacy Study of GSK Biologicals' Quadrivalent Influenza Vaccine, GSK2282512A, (FLU Q-QIV) When Administered in Children
Brief Title: A Study to Evaluate the Efficacy of GSK Biologicals' Influenza Vaccine in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 114541
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FluLaval® Quadrivalent Group (Experimental): Subjects between 3 and 8 years of age at the time of first vaccination received, if primed, 1 dose of FluLaval® Quadrivalent vaccine at Day 0 and, if unprimed, 2 doses of FluLaval® Quadrivalent vaccine at Days 0 and 28. The vaccine was administered intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: FluLaval® Quadrivalent
- Havrix Group (Active Comparator): Subjects between 3 and 8 years of age at the time of first vaccination received, if primed, 1 dose of Havrix™ vaccine at Day 0 and, if unprimed, 2 doses of Havrix™ vaccine at Days 0 and 28. The vaccine was administered intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Havrix™

INTERVENTIONS:
Biological: FluLaval® Quadrivalent — One intramuscular dose for primed subjects. Two intramuscular doses for unprimed subjects.
  Other Names: Quadrivalent seasonal influenza vaccine GSK2282512A
  Arms: FluLaval® Quadrivalent Group
Biological: Havrix™ — Two intramuscular doses for primed subjects. Three intramuscular doses for unprimed subjects.
  Arms: Havrix Group

SUMMARY:
This study is designed to test the efficacy of an investigational influenza vaccine, in children compared to Havrix®, a licensed Hepatitis A virus vaccine.

This study will also evaluate the immunogenicity and safety of the investigational vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s) or legally acceptable representative(s) can and will comply with the requirements of the protocol.
* A male or female child aged between 3 and 8 years inclusive at the time of the first vaccination; children are eligible regardless of history of administration of influenza vaccine in a previous season. However, subjects who have received any seasonal or pandemic influenza vaccine within 6 months preceding the first dose of study vaccine will not be enrolled.
* Written informed consent obtained from the subject/from the parent(s)/legally acceptable representative(s) of the subject.
* Written assent obtained from the subject if/as required by local regulations.
* Subjects in stable health as determined by investigator's clinical examination and assessment of subjects' medical history.
* Access to a consistent means of telephone contact

Exclusion Criteria:

* Child in care.
* Use of an investigational or non-registered product other than the study vaccines within 30 days before study vaccination or planned use during study period. Routine registered childhood vaccinations are permitted.
* Prior receipt of any seasonal or pandemic influenza vaccine within 6 months preceding the first dose of study vaccine, or planned use of such vaccines during the study period. Prior receipt of more than one dose of a licensed hepatitis A vaccine, with the first dose administered at >=12 months of age.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* History of Guillain-Barre syndrome within 6 weeks of receipt of prior influenza virus vaccine.
* Any known or suspected allergy to any constituent of influenza vaccines ; a history of anaphylactic-type reaction to constituent of vaccine; or a history of severe adverse reaction to a previous influenza vaccine.
* Fever at the time of enrolment.
* Acute disease at the time of enrolment.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Ongoing aspirin therapy.
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5220 (Actual)
Dates: Start 2010-12-09; Primary Completion 2012-01-09 (Actual); Study Completion 2012-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- GSK Investigational Site, Dhaka, Bangladesh
- GSK Investigational Site, Santo Domingo, Dominican Republic
- GSK Investigational Site, Tegucigalpa, Honduras
- GSK Investigational Site, Beirut, Lebanon
- GSK Investigational Site, Panama City, Panama
- Philippines (2):
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Dasmariñas, Cavite
- GSK Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Jain VK, Rivera L, Zaman K, Espos RA Jr, Sirivichayakul C, Quiambao BP, Rivera-Medina DM, Kerdpanich P, Ceyhan M, Dinleyici EC, Cravioto A, Yunus M, Chanthavanich P, Limkittikul K, Kurugol Z, Alhan E, Caplanusi A, Durviaux S, Boutet P, Ofori-Anyinam O, Chandrasekaran V, Dbaibo G, Innis BL. Vaccine for prevention of mild and moderate-to-severe influenza in children. N Engl J Med. 2013 Dec 26;369(26):2481-91. doi: 10.1056/NEJMoa1215817. Epub 2013 Dec 11. PMID 24328444
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114541 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114541 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114541 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114541 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114541 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114541 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114541 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 5168 subjects have been enrolled in this study. Primed subjects had received at least 1 dose of an influenza A (H1N1) 2009 monovalent vaccine and had received 2 doses of seasonal influenza vaccine. Unprimed subjects had not received any influenza A (H1N1) 2009 monovalent vaccine or seasonal influenza vaccine.
Pre-assignment Details: The duration of the study was approximately 4-8 weeks to complete enrolment, with at least six months extended safety follow-up (ESFU) after first vaccination, and lasted until the end of the influenza like illness (ILI) surveillance period.
Period: Overall Study
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Started | 2584 | 2584
Completed | 2481 | 2464
Not Completed | 103 | 120
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 61 | 64
Not completed — Lost to Follow-up | 27 | 31
Not completed — Other | 14 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group | Total
Number analyzed (Participants) | 2584 | 2584 | 5168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.4 (1.66) | 5.4 (1.65) | 5.4 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1251 | 1245 | 2496
  Male | 1333 | 1339 | 2672

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least One Confirmed Occurrence of Influenza A or B.
Description: To confirm influenza A and/or B disease, a positive reverse transcriptase polymerase chain reaction (RT-PCR) result for influenza A or B virus from a nose and throat swab obtained concurrently with an influenza like illness (ILI) was required. ILI was defined as the presence of an oral or axillary temperature ≥ 37.8 degrees Celsius (°C) in the presence of at least one of the following symptoms on the same day: cough, sore throat, runny nose or nasal congestion.
Time Frame: From Day 14 to Day 180
Population: The analysis was performed on the According-To-Protocol cohort for efficacy - Time to event, which included all eligible subjects who met all inclusion criteria and no exclusion criteria, followed their study treatment assignment and were successfully contacted at least once after the first vaccination.
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2379 | 2398
subjects | 58 | 128

2. Secondary Outcome: Number of Subjects Reporting at Least One Moderate to Severe Occurrence of Influenza A or B.
Description: To confirm influenza A and/or B disease moderate to severe cases, a positive RT-PCR result for influenza A or B virus from a nose and throat swab obtained concurrently with an ILI was required. Moderate to severe influenza was defined as RT-PCR-confirmed ILI with:
  * Fever >39°C, and/or at least one of the following manifestations,
  * Physician-verified shortness of breath, pulmonary congestion, pneumonia, bronchiolitis, bronchitis, wheezing, croup, or acute otitis media, and/or one of the following,
  * Physician-diagnosed serious extra-pulmonary complication of influenza, including myositis, encephalitis, seizure, or myocarditis
Time Frame: From Day 14 to Day 180
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2379 | 2398
subjects | 14 | 52

3. Secondary Outcome: Number of Subjects Reporting at Least One Culture Confirmed Occurrence of Influenza A or B Due to Antigenically Matched Strain.
Description: To confirm influenza A and/or B disease due to antigenically matched strain, a positive reverse transcriptase polymerase chain reaction (RT-PCR) result for influenza A or B virus from a nose and throat swab obtained concurrently with an influenza like illness (ILI) was required. ILI was defined as the presence of an oral or axillary temperature ≥ 37.8 degrees Celsius (°C) in the presence of at least one of the following symptoms on the same day: cough, sore throat, runny nose or nasal congestion.
Time Frame: From Day 14 to Day 180
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2379 | 2398
subjects | 31 | 56

4. Secondary Outcome: Number of Subjects Reporting at Least One Culture Confirmed Occurrence of Influenza A or B Due to Any Strain.
Description: To confirm influenza A and/or B disease due to any strain, a positive reverse transcriptase polymerase chain reaction (RT-PCR) result for influenza A or B virus from a nose and throat swab obtained concurrently with an influenza like illness (ILI) was required. ILI was defined as the presence of an oral or axillary temperature ≥ 37.8 degrees Celsius (°C) in the presence of at least one of the following symptoms on the same day: cough, sore throat, runny nose or nasal congestion.
Time Frame: From Day 14 to Day 180
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2379 | 2398
subjects | 50 | 112

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was the seropositivity cut-off of 1:10. The 4 influenza strains assessed were the Flu A/California/7/09 (H1N1), Flu A/Victoria/210/09 (H3N2), FluB/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: At Day 0 [PRE] and 28 days post vaccination (Day 28 for primed subjects and day 56 for unprimed subjects) [POST]
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects (those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity outcome measure were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 457 | 122
titers
  H1N1, PRE [N=457;117] | 15.3 [13.6 to 17.3] | 16.1 [12.6 to 20.5]
  H1N1, POST [N=457;121] | 318.8 [291.0 to 349.2] | 16.1 [12.8 to 20.2]
  H3N2, PRE [N=457;117] | 24.3 [21.9 to 27.0] | 28.6 [23.5 to 34.8]
  H3N2, POST [N=457;122] | 264.7 [244.3 to 286.8] | 30.3 [24.8 to 36.9]
  Victoria, PRE [N=457;117] | 13.7 [12.2 to 15.4] | 15.6 [12.2 to 20.1]
  Victoria, POST [N=457;120] | 239.9 [214.6 to 268.2] | 17.8 [13.7 to 23.1]
  Yamagata, PRE [N=457;117] | 16.2 [14.3 to 18.4] | 18.8 [14.4 to 24.5]
  Yamagata, POST [N=457;117] | 361.5 [330.7 to 395.3] | 19.2 [14.9 to 24.7]

6. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer. The 4 influenza strains assessed were the Flu A/California/7/09 (H1N1), Flu A/Victoria/210/09 (H3N2), FluB/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: At 28 days post vaccination (Day 28 for primed subjects and day 56 for unprimed subjects) [POST]
Population: as for outcome 5
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 457 | 117
subjects
  H1N1, POST | 438 | 1
  H3N2, POST | 385 | 2
  Victoria, POST | 425 | 3
  Yamagata, POST | 435 | 1

7. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 4 influenza strains assessed were the Flu A/California/7/09 (H1N1), Flu A/Victoria/210/09 (H3N2), FluB/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: At Day 0 [PRE] and 28 days post vaccination (Day 28 for primed subjects and day 56 for unprimed subjects) [POST]
Population: as for outcome 5
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 457 | 122
subjects
  H1N1, PRE [N=457;117] | 151 | 37
  H1N1, POST [N=457;121] | 451 | 39
  H3N2, PRE [N=457;117] | 205 | 63
  H3N2, POST [N=457;122] | 445 | 63
  Victoria, PRE [N=457;117] | 127 | 35
  Victoria, POST [N=457;120] | 443 | 38
  Yamagata, PRE [N=457;117] | 159 | 45
  Yamagata, POST [N=457;117] | 452 | 45

8. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 4 influenza strains assessed were the Flu A/California/7/09 (H1N1), Flu A/Victoria/210/09 (H3N2), FluB/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: At 28 days post vaccination (Day 28 for primed subjects and day 56 for unprimed subjects) [POST]
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: fold increase
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 457 | 117
fold increase
  H1N1, POST | 20.8 [19.0 to 22.8] | 1.0 [0.9 to 1.1]
  H3N2, POST | 10.9 [9.8 to 12.1] | 1.0 [0.9 to 1.2]
  Victoria, POST | 17.5 [16.0 to 19.1] | 1.1 [1.0 to 1.3]
  Yamagata, POST | 22.3 [20.1 to 24.8] | 1.0 [1.0 to 1.1]

9. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against Each of the 4 Vaccine Strains
Description: HI antibody titres were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Victoria/210/09 (H3N2), Flu B/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: On Day 0 and at least 6 months after first vaccination (Month 6)
Population: The ATP Cohort for persistence included, in terms of antibody response measured by the HI assay, all evaluable subjects for whom data concerning immunogenicity outcome measure were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 444 | 112
Titer
  H1N1, PRE [N=444;112] | 15.5 [13.8 to 17.6] | 16.5 [12.9 to 21.2]
  H1N1, POST [N=444;112] | 138.6 [122.6 to 156.6] | 23.2 [17.9 to 30.1]
  H3N2, PRE [N=444;112] | 24.6 [22.1 to 27.4] | 29.1 [23.8 to 35.5]
  H3N2, POST [N=443;112] | 136.5 [124.3 to 149.9] | 43.6 [34.9 to 54.5]
  Victoria, PRE [N=444;112] | 13.7 [12.2 to 15.4] | 15.1 [11.8 to 19.5]
  Victoria, POST [N=443;112] | 110.2 [97.1 to 125.0] | 19.7 [15.0 to 25.8]
  Yamagata, PRE [N=444;112] | 16.1 [14.2 to 18.4] | 18.7 [14.3 to 24.6]
  Yamagata, POST [N=444;112] | 157.0 [143.1 to 172.3] | 21.8 [16.5 to 28.9]

10. Secondary Outcome: Number of Seroconverted Subjects for HI Antibody Titers Against Each of the 4 Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/California/7/09 (H1N1), Flu A/Victoria/210/09 (H3N2), FluB/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: At least 6 months after first vaccination (Month 6)
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 444 | 112
Subjects
  H1N1, POST [N=444;112] | 349 | 9
  H3N2, POST [N=443;112] | 290 | 10
  Victoria, POST [N=443;112] | 323 | 12
  Yamagata, POST [N=444;112] | 354 | 8

11. Secondary Outcome: Number of Seroprotected Subjects for HI Antibody Titers Against Each of the 4 Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/California/7/09 (H1N1), Flu A/Victoria/210/09 (H3N2), FluB/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: At Day 0 and at least 6 months after first vaccination (Month 6)
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 444 | 112
Subjects
  H1N1, PRE [N=444;112] | 148 | 36
  H1N1, POST [N=444;112] | 383 | 49
  H3N2, PRE [N=444;112] | 204 | 60
  H3N2, POST [N=443;112] | 412 | 71
  Victoria, PRE [N=444;112] | 123 | 32
  Victoria, POST [N=443;112] | 374 | 39
  Yamagata, PRE [N=444;112] | 153 | 43
  Yamagata, POST [N=444;112] | 427 | 49

12. Secondary Outcome: Seroconversion Factors for HI Antibodies Against 4 Strains of Influenza Disease.
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The 4 influenza strains assessed were the Flu A/California/7/09 (H1N1), Flu A/Victoria/210/09 (H3N2), FluB/Brisbane/60/08 (Victoria) and Flu B/Florida/4/06 (Yamagata).
Time Frame: At least 6 months after first vaccination (Month 6)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 444 | 112
Fold increase
  H1N1, POST [N=444;112] | 8.9 [8.1 to 9.8] | 1.4 [1.2 to 1.6]
  H3N2, POST [N=443;112] | 5.5 [5.0 to 6.1] | 1.5 [1.2 to 1.8]
  Victoria, POST [N=443;112 | 8.0 [7.3 to 8.9] | 1.3 [1.1 to 1.6]
  Yamagata, POST [N=444;112] | 9.7 [8.7 to 10.8] | 1.2 [1.0 to 1.4]

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling at the injection site. Any = Incidence of a particular symptom regardless of intensity grade. Grade 3 pain = Cried when limb was moved/spontaneously painful for subjects < 5 years of age or significant pain at rest that prevented normal, everyday activities for subjects ≥ 5 years of age. Grade 3 redness/swelling = Redness/swelling above 100 millimeters (mm) of the injection site. All solicited local symptoms were considered related to vaccination.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and with the symptom sheet completed.
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2546 | 2551
subjects
  Any Pain | 1215 | 888
  Grade 3 Pain | 36 | 20
  Any Redness | 17 | 5
  Grade 3 Redness | 0 | 0
  Any Swelling | 46 | 10
  Grade 3 Swelling | 0 | 0

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms in Subjects Below 5 Years of Age.
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature. Any = Occurrence of any solicited general symptom regardless of intensity grade and relation to vaccination. Any temperature = Axillary temperature ≥ 38.0 °C. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irritability = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = not eating at all. Related = General symptom assessed by the investigator as causally related to the study vaccination. Grade 3 temperature = Axillary temperature ≥ 39.0°C.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination
Population: as for outcome 13
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 899 | 896
subjects
  Any Drowsiness | 100 | 93
  Grade 3 Drowsiness | 5 | 4
  Related Drowsiness | 57 | 61
  Any Irritability | 102 | 91
  Grade 3 Irritability | 5 | 4
  Related Irritability | 60 | 59
  Any Loss of appetite | 119 | 120
  Grade 3 Loss of appetite | 6 | 7
  Related Loss of appetite | 55 | 61
  Any Temperature | 74 | 74
  Grade 3 Temperature | 21 | 18
  Related Temperature | 35 | 35

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms in Subjects of 5 Years of Age and Above.
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (Gastro.), headache, joint pain at other location (Joint pain), muscle aches, shivering and temperature. Any = Occurrence of any solicited general symptom regardless of intensity grade or relation to vaccination. Any temperature = Axillary temperature ≥ 38.0 °C. Grade 3 symptom = Symptom that prevented normal activity. Related = Symptom assessed by the investigator as causally related to the vaccination. Grade 3 temperature = Axillary temperature ≥ 39.0°C.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination
Population: as for outcome 13
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 1648 | 1654
subjects
  Any Fatigue | 188 | 145
  Grade 3 Fatigue | 1 | 6
  Related Fatigue | 101 | 78
  Any Gastro. | 133 | 146
  Grade 3 Gastro. | 9 | 9
  Related Gastro. | 68 | 54
  Any Headache | 243 | 217
  Grade 3 Headache | 9 | 14
  Related Headache | 154 | 125
  Any Joint pain | 143 | 93
  Grade 3 Joint pain | 3 | 2
  Related Joint pain | 98 | 54
  Any Muscle aches | 257 | 194
  Grade 3 Muscle aches | 3 | 5
  Related Muscle aches | 162 | 109
  Any Shivering | 63 | 59
  Grade 3 Shivering | 2 | 2
  Related Shivering | 32 | 26
  Any Temperature | 72 | 82
  Grade 3 Temperature | 21 | 17
  Related Temperature | 46 | 37

16. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = Any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = Unsolicited AE that prevented normal activity. Related = Unsolicited AE assessed by the investigator as causally related to the vaccination.
Time Frame: During the 28-day (Days 0-27) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2584 | 2584
subjects
  Any unsolicited AE(s) | 843 | 855
  Grade 3 unsolicited AE(s) | 25 | 20
  Related unsolicited AE(s) | 30 | 37

17. Secondary Outcome: Number of Subjects With Any and Related Medically Attended Adverse Events (MAEs).
Description: MAEs were defined as AEs that resulted in medical attention (defined as hospitalization, an emergency room visit or a visit to or from medical personnel for any reason). Any = Any MAE regardless of intensity or relationship to vaccination. Related = MAE assessed by the investigator as causally related to the vaccination.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: as for outcome 16
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2584 | 2584
subjects
  Any MAE(s) | 792 | 749
  Related MAE(s) | 6 | 13

18. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs).
Description: pIMDs were defined as a subset of AEs that included both clearly autoimmune diseases (AID) and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Any = Any pIMD(s) regardless of intensity or relationship to vaccination. Related = pIMDs assessed by the investigator as causally related to the vaccination.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: as for outcome 16
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2584 | 2584
subjects
  Any pIMD(s) | 0 | 1
  Related pIMD(s) | 0 | 0

19. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Any = Any SAE(s) regardless of intensity or relationship to vaccination. Related = SAEs assessed by the investigator as causally related to the vaccination.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: as for outcome 16
Measure: Number; unit: subjects
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Number analyzed (Participants) | 2584 | 2584
subjects
  Any SAE(s) | 36 | 24
  Related SAE(s) | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs: during the entire study period (Day 0-Day 180); Unsolicited AEs: during the 28-day (Day 0-Day 27) follow-up period after vaccination; Solicited local/general symptoms: during the 7-day (Day 0-Day 6) follow-up period after any vaccination.
Description: For the systematically assessed other non-serious AEs, the number of participants at risk included those from Total Vaccinated cohort whose symptom sheet had been completed.
Arm/Group | FluLaval® Quadrivalent Group | Havrix Group
Serious Adverse Events (participants affected / at risk) | 36/2584 | 24/2584
Other Adverse Events (participants affected / at risk) | 1215/2584 | 1297/2584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FluLaval® Quadrivalent Group (N=2584) | Havrix Group (N=2584)
Gastroenteritis (Infections and infestations) | 6 | 3
Pneumonia (Infections and infestations) | 4 | 3
Animal bite (Injury, poisoning and procedural complications) | 3 | 1
Dengue fever (Infections and infestations) | 1 | 3
Bronchopneumonia (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 0
Amoebiasis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0
Convulsion (Nervous system disorders) | 1 | 1
Drowning (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Amoebic dysentery (Infections and infestations) | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Croup infectious (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Herpangina (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Optic nerve glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Visceral leishmaniasis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | FluLaval® Quadrivalent Group (N=2584) | Havrix Group (N=2584)
Nasopharyngitis (Infections and infestations) | 213 | 231
Cough (Respiratory, thoracic and mediastinal disorders) | 145 | 137
Pain (General disorders) | 1215/2546 | 888/2551
Drowsiness (General disorders) | 100/899 | 93/896 — Symptom reported for subjects below 5 years of age.
Irritability (General disorders) | 102/899 | 91/896 — Symptom reported for subjects below 5 years of age.
Loss of appetite (General disorders) | 119/899 | 120/896 — Symptom reported for subjects below 5 years of age.
Temperature (General disorders) | 74/899 | 74/896 — Symptom reported for subjects below 5 years of age.
Fatigue (General disorders) | 188/1648 | 145/1654 — Symptom reported for subjects of 5 years of age and above
Gastro. (General disorders) | 133/1648 | 146/1654 — Symptom reported for subjects of 5 years of age and above
Headache (General disorders) | 243/1648 | 217/1654 — Symptom reported for subjects of 5 years of age and above
Joint pain (General disorders) | 143/1648 | 93/1654 — Symptom reported for subjects of 5 years of age and above
Muscle aches (General disorders) | 257/1648 | 194/1654 — Symptom reported for subjects of 5 years of age and above

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.